CLINICAL TRIAL: NCT01058148
Title: A Comparison Study of Two Community Outreach-Based Approaches to Increase Participation of Women Living in the Mississippi Delta in Cervical Cancer Screening
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910036; 10-C-N036
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-13

CONDITIONS: Cervical Intraepithelial Neoplasia; Human Papillomavirus
Keywords: Cervical Cancer Screening; Cervical Precancer; Self-Collection; Cytology; Human Papilloma Virus (HPV)
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* The Mississippi Delta (which includes the counties along the Mississippi River) is one of the poorest areas in the United States. Women living in the Mississippi Delta have disproportionately high rates of cervical cancer, but they are unlikely to come to clinics except perhaps for giving birth, years before they are diagnosed with cancer.
* To improve rates of screening, researchers are attempting an outreach study to see whether under-screened women, if approached by door-to-door recruitment, would get screened by one of two methods (home-based self-collection and testing, or a clinic exam) and which method they would prefer.

Objectives:

- To assess/measure increased participation of under-screened women living in the Mississippi Delta in cervical cancer screening by offering women the opportunity to get screened by one of two possible community outreach-based cervical cancer screening modalities, self-collection and HPV testing or clinic-based cytology screening, the current standard of care.

Eligibility:

- Women between 26 and 65 years of age, who are not pregnant currently or in the past 8 weeks, have an intact cervix, have no history of cancer, and have not been screened for cervical cancer in the past 3 years.

Design:

* Researchers will recruit participants on a door-to-door basis. Researchers will recruit all eligible women within a household. Recruitment will be done only during daylight hours but at the end of the working day to maximize the chances of finding women at home.
* Eligible women willing to participate will complete a questionnaire with demographic and medical information.
* Participants will be asked to choose the screening method of their preference. If they choose self-collection with HPV testing, they will be given a self-collection kit and asked to perform the self-collection and return the kit within 1 month. Participants who choose to have cytology screening will be provided with the phone number and location of the local health department clinic and will be encouraged to schedule their screening within the following month.
* Women who do not complete their participation within 1 month will be considered noncompliant with their chosen intervention. Researchers will re-contact noncompliant women to offer them participation in the study, including permitting them to refuse to participate or to choose the alternative intervention....

DETAILED DESCRIPTION:
We have been conducting a study of self-collected cervicovaginal specimens and carcinogenic human papillomavirus (HPV) DNA testing for cervical cancer screening of women living in the Mississippi Delta, who have disproportionately high rates of cervical cancer. To date, we have noted high levels of participation as well as high percentages of completion and return of the home self-collection. Although we have recruited some under-screened women into our study, it was clinic-based (i.e., under-screened women were still required to come to the health department clinic), using Mississippi State Department of Health district clinics. In reality, women who get cervical cancer in the Mississippi Delta are unlikely to come to clinics except perhaps for giving birth, years before they are diagnosed with cancer. Thus, as an ancillary study to our work in Mississippi, we are proposing an outreach study to determine whether under-screened women, if approached via door-to-door recruitment, would participate (get screened) by one of two community outreach-based cervical cancer screening modalities, home-based self-collection and HPV testing or clinic-based cytology screening, and which of the two modalities they prefer. We will recruit door-to-door 400 under-screened, eligible women aged 26-65 years living in the Mississippi Delta. Consenting, eligible women will be given a choice of taking and using a self-collection kit on their own or coming to the local Health Department clinic for cervical cytology screening. Under the assumption that only 5% of this under-screened population would choose to undergo screening without intervention, recruitment of 400 women into the study will permit us to detect a 2-fold increase in participation in screening (defined as completing screening) with 90% power (alpha = 0.05). In this scenario, we will be able to detect with 90% power (alpha = 0.05) a 25% preference for one of the screening methods (75% vs. 50% (no preference)).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Women who are age 26-65 years, not pregnant currently or in the past 8 weeks, who have an intact cervix, no history of cancer, have not been screened for cervical cancer in the last 3 years, and able and competent to provide informed consent will be considered eligible for the study.

EXCLUSION CRITERIA:

* Women under 26 or over 65 years of age.
* Pregnant women or women who have given birth to a child in the past 8 weeks. To insure women included in the study are not pregnant, we will ask women during the consenting process if they are pregnant or gave recently given birth. Women who answer yes for either query will be excluded.
* Women who have had a total hysterectomy.
* History of cervical cancer
* Screened for cervical cancer in the last 3 years.
* Other reasons to exclude women include the inability to speak English, the appearance of mental incompetence, or refusal to participate or sign the informed consent form.

Ages: 26 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-12-22; Study Completion 2011-04-13

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Cuzick J, Clavel C, Petry KU, Meijer CJ, Hoyer H, Ratnam S, Szarewski A, Birembaut P, Kulasingam S, Sasieni P, Iftner T. Overview of the European and North American studies on HPV testing in primary cervical cancer screening. Int J Cancer. 2006 Sep 1;119(5):1095-101. doi: 10.1002/ijc.21955. PMID 16586444
- [Background] Dillner J, Rebolj M, Birembaut P, Petry KU, Szarewski A, Munk C, de Sanjose S, Naucler P, Lloveras B, Kjaer S, Cuzick J, van Ballegooijen M, Clavel C, Iftner T; Joint European Cohort Study. Long term predictive values of cytology and human papillomavirus testing in cervical cancer screening: joint European cohort study. BMJ. 2008 Oct 13;337:a1754. doi: 10.1136/bmj.a1754. PMID 18852164